CLINICAL TRIAL: NCT03293550
Title: The Association Between Minor Brain Injuries and Level of Anesthesia Detected by a New EEG Based Tool, to Delirium and Post-operative Cognitive Dysfunction After Cardiac and Non-cardiac Surgery - a Proof of Concept Study
Brief Title: Can a New EEG Based Tool Predict Post-operative Delirium and Cognitive Dysfunction?
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Neuroindex Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 185-17 rambam-CTIL
Record Dates: First submitted 2017-08-31; First posted 2017-09-26 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Delirium; Cognitive Dysfunction
MeSH Terms: conditions — Delirium; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients over 65 years undergoing elective surgery: patients over 65 years undergoing elective cardiac surgery or elective hip or knee surgery

SUMMARY:
As the population ages and medical progress is made, many elderly patients that previously would not have been candidates for surgery are now undergoing operations. In this group of older patients, brain dysfunction after anesthesia and surgery is well recognized and categorized into two distinct clinical entities; Post-operative cognitive delirium (POD) and post-operative cognitive dysfunction (POCD).

Delirium is an acute and fluctuating deterioration in attention accompanied by either a change in cognition or arousal and is often diagnosed by criteria established in the Confusion Assessment Method (CAM). Delirium can present as hypoactive (decreased alertness, motor activity and anhedonia), as hyperactive (agitated and combative) or as mixed forms. Age and the type of operation are the major risk factors.

Post-operative cognitive dysfunction (POCD) is a term used to describe subtle changes in cognition, such as memory and executive function. The most commonly seen problems are memory impairment and impaired performance on intellectual tasks. In severe cases, it can lead to inability to perform daily living functions. It was previously found that the presence of cognitive dysfunction 3 months after non-cardiac surgery was associated with an increased mortality. The mechanisms leading to cognitive impairment after anesthesia and surgery are not yet fully clear. The risk factors are related to patient characteristics, type of operation and anesthetic management.

Despite its limitations over-anesthesia as monitored by BIS was at-least correlative with POD. Therefore it is hopeful that an even more precise evaluation of the level of anesthesia will improve POD prediction (and thereby prevention) even further.

On the other hand the measure of depth of anesthesia by itself does not provide sufficient prediction for POCD. In POCD a major role has been assigned to hippocampal damage.

The investigators have recently demonstrated that temporary hippocampal interruptions are manifested by interhemispheric desynchronization, which are recognized by our new algorithm, which monitors electrophysiological markers of attention and of perception.

The investigators have developed a unique algorithm for analyzing EEG based on the concept of monitoring perception and attention and their interhemispheric synchronization.

The aims of this proof of concept study are: (i) to find-out whether interhemispheric desynchronization of attentional processes is associated with POCD; (ii) to find out whether the level of anesthesia, is linked primary to POD and secondary to POCD.

DETAILED DESCRIPTION:
As the population ages and medical progress is made, many elderly patients that previously would not have been candidates for surgery are now undergoing operations. In this group of older patients, brain dysfunction after anesthesia and surgery is well recognized and categorized into two distinct clinical entities; Post-operative cognitive delirium (POD) and post-operative cognitive dysfunction (POCD).

Delirium is an acute and fluctuating deterioration in attention accompanied by either a change in cognition or arousal and is often diagnosed by criteria established in the Confusion Assessment Method (CAM). Delirium can present as hypoactive (decreased alertness, motor activity and anhedonia), as hyperactive (agitated and combative) or as mixed forms. Age and the type of operation are the major risk factors.

Post-operative cognitive dysfunction (POCD) is a term used to describe subtle changes in cognition, such as memory and executive function. The most commonly seen problems are memory impairment and impaired performance on intellectual tasks. In severe cases, it can lead to inability to perform daily living functions. The reported incidence figures for postoperative cognitive dysfunction vary depending on the group of patients studied, the definition of POCD used, the tests used to establish the diagnosis and their statistical evaluation, the timing of testing, and the choice of control group. The diagnosis of POCD relies on the use of neuropsychological tests, including; visual verbal learning test, based on Rey's auditive recall of words, the concept shifting test, based on the trail- making test from Halstead and Reitan's neuropsychological test battery, the Stroop color word interference test , the letter-digit coding, based on the symbol-digit substitution task from the Wechsler adult intelligence scale and the four boxes test. In a large prospective multicenter cohort study, it was found that the presence of cognitive dysfunction 3 months after noncardiac surgery was associated with an increased mortality. Furthermore, patients with cognitive decline at 1 week had an increased risk of leaving the labor market prematurely and a higher prevalence of time receiving social transfer payments. The mechanisms leading to cognitive impairment after anesthesia and surgery are not yet fully clear. The risk factors for developing POCD are related to patient characteristics, type of operation and anesthetic management.

Cardiovascular, respiratory, hepatic, and renal insufficiency are all associated with impaired brain performance. It is theoretically obvious that an adequate intraoperative oxygen supply for all vital organs is essential if postoperative cerebral dysfunction is to be avoided. Casai et al found that brain desaturation (rSO2 decrease <75% of baseline) occurred in 40% of elderly patients after noncardiac surgery, and the cerebral desaturation was linked with a high incidence of POCD. A recent systematic review shows that reductions in cerebral oxygen saturation (rSO2) during cardiac surgery may indicate CPB cannula malposition, particularly during aortic surgery. However, only weak evidence links low rSO2 during cardiac surgery to POCD.

POCD is a well-recognized clinical phenomenon of multifactorial origin; emboli, hypoperfusion, inflammation, and patient's preoperative cerebral dysfunction Meticulous surgical and anesthesiological techniques are important for preventing complications and keeping the risk of POCD to a minimum.

The EEG is an electrophysiological monitoring method used to record electrical activity of the brain, including normal and abnormal activity. In recent years, numerous clinical studies were performed to evaluate whether the use in intraoperative electroencephalography (EEG) to control the depth of anesthesia has any effect on POCD.

Recently it was confirmed that intraoperative neuro-monitoring for depth of anesthesia is associated with a lower incidence of delirium. However it is unrelated to the incidence of POCD. The most common available monitor for depth of anesthesia is the Bispectral index, developed more than 20 years ago. The device's output is based on electroencephalographic (EEG) signals from the frontal lobe (monitors brain activity) in combination with electromyographic (EMG) waves (monitors muscle activity). The BIS produces a number ranging from 0 -100, which matches the patient's level of consciousness (awake, sedated or unconscious) under GA. There are two main problems with the BIS device: (1) It analyzes EEG and EMG with no ability to differentiate the neuronal activity from the muscle activity. Thus, when neuromuscular blocking drugs (NMBDs) are used, scores produced by the BIS are influenced by the lack of muscle activity, and mistakenly indicate a state of unconsciousness (lack of neuronal activity) even if no hypnotic medications were used, and (2) The BIS is based solely on frontal electrodes and does not monitor posterior activity. Thus, anesthetic medications with more posterior effect (such as ketamine) receive a false score by the BIS device. Accordingly, the BIS system might be better used as a means of tracking specific anesthetic medications and not as a universal means for monitoring unconsciousness.

Despite its limitations over-anesthesia as monitored by BIS was at-least correlative with POD (but not with POCD). Therefore it is hopeful that an even more precise evaluation of the level of anesthesia will improve POD prediction (and thereby prevention) even further. On the other hand the measure of depth of anesthesia by itself does not provide sufficient prediction for POCD. In POCD a major role has been assigned to hippocampal damage.

The investigators have recently demonstrated that temporary hippocampal interruptions are manifested by interhemispheric desynchronization, which are recognized by our new algorithm, which monitors electrophysiological markers of attention and of perception. This algorithm was based on a previous set of studies, which showed the ability to decompose the entire multi-electrode EEG/ERP sample to a superposition of attention and perception processes, spread in space (over the scalp) and time (hundreds of milliseconds). Our algorithm is unique in the ability to extract the needed perceptual and attentional information indicating depth of anesthesia and hemispheric damage (manifested by interhemispheric desynchronization) in real time every 30 seconds and with a minimal electrodes setup, comprised of 6 electrodes.

The aims of this proof of concept study are: (i) to find-out whether interhemispheric desynchronization of attentional processes is associated with POCD; (ii) to find out whether the level of anesthesia, is linked primary to POD and secondary to POCD. For both purposes the investigators use a novel EEG algorithm based on the concept of monitoring perception and attention and their interhemispheric synchronization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 65 years or older undergoing elective cardiac surgery (CABG or valve replacement) or hip/knee replacement.

Exclusion Criteria:any of the following criteria;

1. inability or refusal to provide informed consent,
2. significant visual impairment so that the pictures of the confusion assessment method could not be interpreted to accurately test to assess delirium,
3. profound dementia or aphasia that interfered with the assessment of delirium,
4. inability to speak Hebrew/ Russian or Arabic so that a language barrier was not confused with postoperative confusion.
5. Any previously documented major neurologic or psychiatric dysfunction

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients 65 years or older, ASA 1-4, undergoing elective cardiac surgery (CABG or valve replacement) or hip/knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-12-31 (Actual); Primary Completion 2020-09-06 (Actual); Study Completion 2020-09-06 (Actual)

PRIMARY OUTCOMES:
Correlation of depth of anesthesia to post operative delirium | The diagnosis of delirium is assessed two hours after the operation, when the patient is fully awake, in the post anesthesia care unit (PACU)
  Correlation of depth of anesthesia, as measured by a new EEG based algorithm, to post operative delirium
Correlation of intra operative EEG changes to early post operative cognitive dysfunction | The diagnosis of cognitive dysfunction is assessed post operative on day 7 and compared to baseline pre surgery cognitive function.
  Correlation of EEG changes as measured by a new EEG based algorithm to post operative cognitive dysfunction
Correlation of intra operative EEG changes to 45 days post operative cognitive dysfunction | The diagnosis of cognitive dysfunction is assessed post operative on day 45 and is compared to baseline pre surgery cognitive function.
  Correlation of EEG changes as measured by a new EEG based algorithm to post operative cognitive dysfunction
Correlation of intra operative EEG changes to late post operative cognitive dysfunction | The diagnosis of cognitive dysfunction is assessed post operative on day 90 and is compared to baseline pre surgery cognitive function.
  Correlation of EEG changes as measured by a new EEG based algorithm to post operative cognitive dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Audisio R, Borozdina A, Cherubini A, Jones C, Kehlet H, MacLullich A, Radtke F, Riese F, Slooter AJ, Veyckemans F, Kramer S, Neuner B, Weiss B, Spies CD. European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium. Eur J Anaesthesiol. 2017 Apr;34(4):192-214. doi: 10.1097/EJA.0000000000000594. PMID 28187050
- [Background] Avidan MS, Zhang L, Burnside BA, Finkel KJ, Searleman AC, Selvidge JA, Saager L, Turner MS, Rao S, Bottros M, Hantler C, Jacobsohn E, Evers AS. Anesthesia awareness and the bispectral index. N Engl J Med. 2008 Mar 13;358(11):1097-108. doi: 10.1056/NEJMoa0707361. PMID 18337600
- [Background] Brown C 4th, Deiner S. Perioperative cognitive protection. Br J Anaesth. 2016 Dec;117(suppl 3):iii52-iii61. doi: 10.1093/bja/aew361. PMID 27940456
- [Background] Casati A, Fanelli G, Pietropaoli P, Proietti R, Tufano R, Montanini S; Collaborative Italian Study Group on Anaesthesia in Elderly Patients; Danelli G, Nuzzi M, Mentegazzi F, Torri G, Martani C, Spreafico E, Fierro G, Pugliese F, De Cosmo G, Aceto P, Servillo G, Monaco F. Monitoring cerebral oxygen saturation in elderly patients undergoing general abdominal surgery: a prospective cohort study. Eur J Anaesthesiol. 2007 Jan;24(1):59-65. doi: 10.1017/S0265021506001025. Epub 2006 Jul 7. PMID 16824246
- [Background] Chan MT, Cheng BC, Lee TM, Gin T; CODA Trial Group. BIS-guided anesthesia decreases postoperative delirium and cognitive decline. J Neurosurg Anesthesiol. 2013 Jan;25(1):33-42. doi: 10.1097/ANA.0b013e3182712fba. PMID 23027226
- [Background] Glass PS, Bloom M, Kearse L, Rosow C, Sebel P, Manberg P. Bispectral analysis measures sedation and memory effects of propofol, midazolam, isoflurane, and alfentanil in healthy volunteers. Anesthesiology. 1997 Apr;86(4):836-47. doi: 10.1097/00000542-199704000-00014. PMID 9105228
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Paredes S, Cortinez L, Contreras V, Silbert B. Post-operative cognitive dysfunction at 3 months in adults after non-cardiac surgery: a qualitative systematic review. Acta Anaesthesiol Scand. 2016 Sep;60(8):1043-58. doi: 10.1111/aas.12724. Epub 2016 Mar 29. PMID 27027720
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Radtke FM, Franck M, Lendner J, Kruger S, Wernecke KD, Spies CD. Monitoring depth of anaesthesia in a randomized trial decreases the rate of postoperative delirium but not postoperative cognitive dysfunction. Br J Anaesth. 2013 Jun;110 Suppl 1:i98-105. doi: 10.1093/bja/aet055. Epub 2013 Mar 28. PMID 23539235
- [Background] Short TG, Campbell D, Leslie K. Response of bispectral index to neuromuscular block in awake volunteers. Br J Anaesth. 2016 May;116(5):725-6. doi: 10.1093/bja/aew089. No abstract available. PMID 27106988
- [Background] Shahaf DB, Shahaf G, Mehta J, Venkatraghavan L. Intracarotid Etomidate Decreases the Interhemispheric Synchronization in Electroencephalogram (EEG) During the Wada Test. J Neurosurg Anesthesiol. 2016 Oct;28(4):341-6. doi: 10.1097/ANA.0000000000000241. PMID 26536542
- [Background] Shahaf G, Fisher T, Aharon-Peretz J, Pratt H. Comprehensive analysis suggests simple processes underlying EEG/ERP - demonstration with the go/no-go paradigm in ADHD. J Neurosci Methods. 2015 Jan 15;239:183-93. doi: 10.1016/j.jneumeth.2014.10.016. Epub 2014 Nov 1. PMID 25445244
- [Background] Shahaf G, Pratt H. Thorough specification of the neurophysiologic processes underlying behavior and of their manifestation in EEG - demonstration with the go/no-go task. Front Hum Neurosci. 2013 Jun 24;7:305. doi: 10.3389/fnhum.2013.00305. eCollection 2013. PMID 23805094
- [Background] Wildes TS, Winter AC, Maybrier HR, Mickle AM, Lenze EJ, Stark S, Lin N, Inouye SK, Schmitt EM, McKinnon SL, Muench MR, Murphy MR, Upadhyayula RT, Fritz BA, Escallier KE, Apakama GP, Emmert DA, Graetz TJ, Stevens TW, Palanca BJ, Hueneke R, Melby S, Torres B, Leung JM, Jacobsohn E, Avidan MS. Protocol for the Electroencephalography Guidance of Anesthesia to Alleviate Geriatric Syndromes (ENGAGES) study: a pragmatic, randomised clinical trial. BMJ Open. 2016 Jun 15;6(6):e011505. doi: 10.1136/bmjopen-2016-011505. PMID 27311914